CLINICAL TRIAL: NCT03774524
Title: Effects of Co-administered Sublingual Misoprostol and Intravenous Tranexamic Acid on Prevention of Postpartum Hemorrhage in Pregnant Women With Twin Pregnancy Undergoing Elective Cesarean Section: A Double-Blind Randomized Clinical Trial
Brief Title: Sublingual Misoprostol and Tranexamic Acid in Pregnant Women With Twin Pregnancy Undergoing Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu / 183/18
Record Dates: First submitted 2018-12-12; First posted 2018-12-13 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Cesarean Section Complications
Keywords: cesarean section; tranexamic acid; postpartum hemorrhage; misoprostol
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Intervention Model Description: A Double-Blind Randomized Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: a double-blinded randomized placebo-controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Misoprostol with TA (Active Comparator): 400 μg of sublingual misoprostol (two tablets) plus 1 gm tranexamic acid in 100 ml saline by iv rout
  Interventions: Drug: Misoprostol; Drug: TA
- Misoprostol with placebo to TA (Active Comparator): 400 μg of sublingual misoprostol (two tablets) plus 110 ml saline by iv rout
  Interventions: Drug: Misoprostol; Drug: placebo to misoprostol
- placebo to Misoprostol with placebo to TA (Placebo Comparator): placebo to misoprostol plus placebo to tranexamic acid
  Interventions: Drug: placebo to misoprostol; Drug: placebo to TA

INTERVENTIONS:
Drug: Misoprostol — 400 μg of sublingual misoprostol
  Other Names: Active Comparator
  Arms: Misoprostol with TA; Misoprostol with placebo to TA
Drug: TA — 1 gm of tranexamic acid in 100 ml saline iv
  Other Names: Active Comparator
  Arms: Misoprostol with TA
Drug: placebo to misoprostol — placebo tablets to misoprostol subligual
  Other Names: Placebo comparator
  Arms: Misoprostol with placebo to TA; placebo to Misoprostol with placebo to TA
Drug: placebo to TA — 110 ml saline iv
  Other Names: placebo comparator
  Arms: placebo to Misoprostol with placebo to TA

SUMMARY:
Purpose to evaluate the effects of sublingual misoprostol with or without intravenous tranexamic acid (TA) in comparison with placebo on reducing post-partum hemorrhage in pregnant women with twin pregnancy undergoing an elective cesarean section.

DETAILED DESCRIPTION:
Uterine atony is the major cause of postpartum hemorrhage (PPH), accounting for up to 80% of PPH cases. PPH is the leading cause of maternal morbidity and mortality worldwide, resulting in up to 28% of maternal deaths. Therefore, inducing a rapid and effective uterine contraction following delivery is an important issue. Risk factors of uterine atony include obesity, White or Hispanic race/ethnicity, polyhydramnios, preeclampsia, anemia, and chorioamnionitis as well as a twin pregnancy.

With the increasingly common use of ovulation induction and assisted reproduction techniques, the incidence of multiple gestation pregnancies has progressively increased. Suzuki et al reported that elective cesarean delivery of twin pregnancy at a gestational age of 37 weeks or greater may increase the risk of blood transfusion. Several uterotonic agents are used to prevent PPH because of uterine atony, including oxytocin, an ergot alkaloid, and prostaglandin. However, there are currently no data to evaluate the efficacy of co-administered Sublingual Misoprostol and Intravenous Tranexamic Acid on prevention of postpartum hemorrhage in pregnant women with twin pregnancy undergoing an elective cesarean. therefore, this study was designed to evaluate and compare these two new therapeutic options in controlling PPH following CS for twin pregnancy

ELIGIBILITY:
Inclusion Criteria:

* women with a multiple term pregnancy undergoing elective cesarean section

Exclusion Criteria:

* single gestation
* placenta praevia and placental abruption
* undergoing cesarean section with general anesthesia
* women undergoing cesarean section at less than 37 weeks of gestation
* with a severe medical disorder
* allergy to tranexamic acid or misoprostol

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women with a multiple term pregnancy undergoing elective cesarean section
Enrollment: 150 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
estimation of intraoperative blood loss (ml) | during the operation
  measure Intraoperative blood loss in ml by gravimetric methods

SECONDARY OUTCOMES:
amount of postoperative blood loss | 6 hours post operative
  measure amount of blood loss post operative in ml by gravimetric methods
number of patient with postpartum hemorrhage | 24 hours post operative
  calculation of the number of the patients with blood loss >1000 ml

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided